CLINICAL TRIAL: NCT05991050
Title: Effect of Whole Body Vibration on Blood Pressure in Obese Postmenopausal Women. A Randomized Controlled Study
Brief Title: Effect of Whole Body Vibration on Blood Pressure in Obese Postmenopausal Women.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 70
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet regimen group (Active Comparator): an energy-restricted diet for 8 weeks. Meal plan that creates an energy deficit of 500 to 1000 Kcal per day less than the individual's average daily intake was suitable for weight reduction.Each post-menopausal woman followed Dietary Approaches to Stop Hypertension (DASH) which : low in total fat, cholesterol, red meat, sweets and sugar containing beverages, emphasize fish, nuts, fruits, vegetables and whole grains and it also rich in Potassium(6900mg), Calcium(1200-1500mg) and Magnesium, as well as vitamins A, C and E.
  Interventions: Dietary Supplement: energy-restricted diet
- whole body vibration group (Active Comparator): For 8 weeks, WBV participants completed 3 supervised training sessions a week. The exercises were consisted of dynamic squats starting from upright position into the assigned degree of knee ﬂexion "squats with 90° knee angle, semi-squats with 120° knee angle" and heel elevation (calf-raise), each exercise was performed for 3 sets and each set consisted of 5 repetitions.
  Interventions: Dietary Supplement: energy-restricted diet; Device: Whole body vibration

INTERVENTIONS:
Dietary Supplement: energy-restricted diet — Meal plan that creates an energy deficit of 500 to 1000 Kcal per day less than the individual's average daily intake was suitable for weight reduction.Each post-menopausal woman followed Dietary Approaches to Stop Hypertension (DASH) which : low in total fat, cholesterol, red meat, sweets and sugar containing beverages, emphasize fish, nuts, fruits, vegetables and whole grains and it also rich in Potassium(6900mg), Calcium(1200-1500mg) and Magnesium, as well as vitamins A, C and E.
Device: Whole body vibration — For 8 weeks, WBV participants completed 3 supervised training sessions a week. The exercises were consisted of dynamic squats starting from upright position into the assigned degree of knee ﬂexion "squats with 90° knee angle, semi-squats with 120° knee angle" and heel elevation (calf-raise), each exercise was performed for 3 sets and each set consisted of 5 repetitions.
  Arms: whole body vibration group

SUMMARY:
All post-menopausal women followed an energy-restricted diet for 8 weeks. Meal plan that creates an energy deficit of 500 to 1000 Kcal per day less than the individual's average daily intake was suitable for weight reduction.Each post-menopausal woman followed Dietary Approaches to Stop Hypertension (DASH) which : low in total fat, cholesterol, red meat, sweets and sugar containing beverages, emphasize fish, nuts, fruits, vegetables and whole grains and it also rich in Potassium(6900mg), Calcium(1200-1500mg) and Magnesium, as well as vitamins A, C and E.Group B (WBV group):

For 8 weeks, WBV participants completed 3 supervised training sessions a week.

DETAILED DESCRIPTION:
I-Group A (control group):

All post-menopausal women followed an energy-restricted diet for 8 weeks. Meal plan that creates an energy deficit of 500 to 1000 Kcal per day less than the individual's average daily intake was suitable for weight reduction.Each post-menopausal woman followed Dietary Approaches to Stop Hypertension (DASH) which : low in total fat, cholesterol, red meat, sweets and sugar containing beverages, emphasize fish, nuts, fruits, vegetables and whole grains and it also rich in Potassium(6900mg), Calcium(1200-1500mg) and Magnesium, as well as vitamins A, C and E.

II-Group B (WBV group):

For 8 weeks, WBV participants completed 3 supervised training sessions a week. Each participant received an explanation of the WBV device and the treatment protocol. Women stood in upright position and hold on handle bar before switching the WBV device at "on" position.

The exercises were consisted of dynamic squats starting from upright position into the assigned degree of knee ﬂexion "squats with 90° knee angle, semi-squats with 120° knee angle" and heel elevation (calf-raise), each exercise was performed for 3 sets and each set consisted of 5 repetitions. All dynamic exercises were performed with slow controlled movements and between each set, there was resting period during which women assumed upright standing position for 1 minute. Total duration of the training session was 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 -65 years
* BMI 30 to 34.99 Kg / m2
* prehypertension and hypertension stage I

Exclusion Criteria:

* systolic blood pressure exceeding 159 mm Hg and diastolic blood pressure exceeding 99 mm Hg,
* diabetic neuropathy disease,
* patients with mental or psychological disorders,
* skin disorders or bleeding disorders, and
* musculoskeletal disorders that limited WBV.

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Blood pressure measurement | before and after 8 weeks of treatment
  The auscultatory method of measuring both systolic and diastolic blood pressure was used with a sphygmomanometer properly calibrated and validated

SECONDARY OUTCOMES:
Anthropometric measurements | before and after 8 weeks of treatment
  using standardized equipment (Weight and height scale). Height of all participants were measured in standing position without footwear. Body mass index was then calculated

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Maged, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No